CLINICAL TRIAL: NCT01581957
Title: A Pilot Study to Evaluate the Effect of a Specific Enteral Formulation Designed to Improve Gastrointestinal Tolerance in the Critically Ill Patient
Brief Title: Pilot Study on Gastro-intestinal (GI) Enteral Nutrition (EN) Tolerance in Intensive Care Unit Patients
Acronym: SPIRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 10.10.CLI
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Critically Ill
Keywords: Enteral nutrition, critically ill patients
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Specific Enteral formulation (Active Comparator)
  Interventions: Other: Specific Enteral Nutrition
- Standard enteral formulation (Placebo Comparator)
  Interventions: Other: Standard Enteral Nutrition

INTERVENTIONS:
Other: Specific Enteral Nutrition — Patients will receive a Specific EN. The caloric target is 25 Kcal/kg/day to be reached on the third day post-initiation of EN (early enteral nutrition).
  Arms: Specific Enteral formulation
Other: Standard Enteral Nutrition — Patients will receive an equivalent volume and caloric intake of standard formulation. The caloric target is 25 Kcal/kg/day to be reached on the third day post-initiation of EN (early enteral nutrition).
  Arms: Standard enteral formulation

SUMMARY:
Specifically designed enteral formulations may improve the gastrointestinal tolerance during early enteral nutrition in the critically ill patient.

This pilot trial will permit testing the design of the full-scale study providing valuable data on the expected effect of the formulation, the variability, thus helping to better estimate the required sample size.

ELIGIBILITY:
Inclusion Criteria:

* Male or female older than 18 years of age
* All ICU patients
* Expected ICU stay superior or equal to 5 days
* Anticipated to receive tube feeding for at least 3 days
* Informed consent obtained from patient or close relative

Exclusion Criteria:

* Contraindication to enteral nutrition or to the placement of an enteral feeding tube
* On enteral nutrition with superior or equal to 75% of caloric goal administered
* Restriction in full intestinal support including protein administration
* Parenteral nutrition of any kind unless due to enteral nutrition intolerance
* History of allergy or intolerance to the study product components (test or control product)
* Currently under therapeutic limitations. Non functional GI tract
* Unwilling or unable to comply with study treatments
* Currently participating or having participated in another clinical, interventional trial during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-12; Primary Completion 2014-02 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Diarrhea-free days during Enteral Nutrition (EN) administration to the patients in the Intensive Care Unit (ICU) | from EN start until end of treatment or ICU discharge (whatever comes first)
  Patients will receive treatment for 10 days maximum
Number of diarrhea events per day during EN administration to the patients in the Intensive Care Unit (ICU) | from EN start until end of treatment or ICU discharge (whatever comes firts)
  Patients will receive treatment for 10 days maximum

SECONDARY OUTCOMES:
Incidence and severity of diarrhea | up to 10 days
  * Number of patients that experienced diarrhea during ICU stay
  * Interruption of EN due to diarrhea
  * Presence/absence of electrolyte and acid-base disturbances secondary to diarrhea
Presence/absence of other abdominal symptoms | up to 10 days
  If present: description of abdominal distension, pain, absence of bowel sounds
Changes in intra-abdominal pressure | up to 10 days
Incidence of nausea, vomiting and regurgitation | up to 10 days
Gastric residual volumes (>500 ml) | up to 10 days
Need to use any drug interfering with the passage of nutrition | up to 10 days
Visual analogue scale for abdominal discomfort | up to 10 days
  Assessed in non-comatose patients
Health Economic burden of Diarrhea during EN administration at ICU | up to 10 days
  * Nurse workload for the management of patients with diarrhea during the EN feeding period in ICU
  * Total cost of diarrhea evaluated for each patient who experienced diarrhea (medications, cleaning material, blankets, etc.)
For blood glucose control | up to 10 days
  * Number of events outside the 4.5 to 10 mmol/l glycaemic range
  * Need for insulin unit administration during exclusive enteral nutrition
  * Need for glucose administration during exclusive enteral nutrition
Time to reach the full caloric goal | up to 10 days
  25 Kcal/kg/day or as determined for each patient with indirect calorimetry
Accumulated daily caloric deficit during 72 hs after start of the study | up to 10 days
  Percentage of cumulative calories delivered vs. prescribed during hospitalization in ICU and accumulated deficit during ICU stay/day (it should be the same)
Need for parenteral nutrition supplementation during ICU stay | up to 10 days
  yes/no, economic impact
Nutritional assessment | up to 10 days
  serum albumin at baseline, 3 days after EN start and at treatment end or at ICU discharge (whatever comes first)
Incidence of secondary infections | up to 10 days
ICU Length of Stay, days on mechanical ventilation during ICU stay (mech. ventilation-free days), hospital LOS (length of stay) | up to 28 days
Microbiota profiling | up to 10 days
  Comprehensive intestinal microbiota profiling by sequencing-based approaches in stool samples collected right before initiation of EN, 3 days after EN start, at treatment end or at ICU discharge (whatever comes first), and at diarrhea episodes
Determination of diarrhea pathogenicity | up to 10 days
  Infections, fecal cultures for pathogens assessed at diarrhea episodes
Safety evaluation (blood sampling) | up to 10 days
  End-point of safety evaluation at baseline, 3 days after EN start and at treatment end or at ICU discharge (whatever comes first), will include: blood cell analysis, hemoglobin, hepatic enzymes and creatinine
AEs (adverse events) / SAEs (serious adverse events) | up to 28 days
  AE and SAE reporting from study start until 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Jakob, Professor, Principal Investigator — Bern University Hospital
Locations (1):
- Department of Intensive Care Medicine. Bern University Hospital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Derived] Jakob SM, Butikofer L, Berger D, Coslovsky M, Takala J. A randomized controlled pilot study to evaluate the effect of an enteral formulation designed to improve gastrointestinal tolerance in the critically ill patient-the SPIRIT trial. Crit Care. 2017 Jun 10;21(1):140. doi: 10.1186/s13054-017-1730-1. PMID 28599662